CLINICAL TRIAL: NCT01099137
Title: The Study About Glucose Lowering Effect of Vildagliptin in Type 2 Diabetes Patients Who Are Uncontrolled With Metformin and a Sulphonylurea
Brief Title: Effect of Vildagliptin in Type 2 Diabetes Treated With Sulphonylurea and Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUBH_ENDO3
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes
Keywords: Diabetes; Vildagliptin; insulin; C-peptide
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Vildagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vildagliptin (Experimental): Vildagliptin will be added to uncontrolled diabetic patients with sulphonylurea and metformin
  Interventions: Drug: Vildagliptin
- Sulphonylurea dose-up (Active Comparator): Sulphonylurea dose will be increased to uncontrolled diabetic patients with sulphonylurea and metformin
  Interventions: Drug: Sulphonylurea dose-up

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50mg twice a day, orally, for 24 weeks
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Sulphonylurea dose-up — glimepiride dose will be increased by 50% to uncontrolled diabetic patients with glimepiride and metformin
  Other Names: Amaryl
  Arms: Sulphonylurea dose-up

SUMMARY:
Dual combination therapy with metformin and sulphonylurea is the most commonly used combination regimen to treat patients with type 2 diabetes. But, treatment with the dual combination therapy is often unsuccessful at achieving glycaemic control in patients with type 2 diabetes. In this setting, use of insulin is often the next therapeutic step.

Recently, dipeptidyl peptidase (DPP)-IV inhibitor is increasingly being used in clinical practice. It is well established that DPP-IV inhibitor improve glycemic control in patients with type 2 diabetes.

But, there have been few studies about the glucose lowering effect of DPP-IV inhibitors (vildagliptin) in Type 2 diabetes patients on the dual combination therapy with a sulfonylurea agent and metformin.The researchers hypothesized that DPP-IV inhibitor as add-on therapy to combination of a sulfonylurea agent and metformin have favorable glucose lowering effect in type 2 diabetic patients. The researchers plan to investigate the change in HbA1C and fasting glucose of 24 weeks treatment with vildagliptin (DPP-IV inhibitor) in combination with a sulfonylurea agent and metformin in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c ≥ 7%
* Age ≥ 18

Exclusion Criteria:

* Contraindication to Vildagliptin
* Pregnant or breast feeding women
* Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
* Chronic hepatitis B or C (except healthy carrier of HBV)
* Liver disease (AST/ALT > 3-fold the upper limit of normal)
* Renal failure (Cr > 2.0)
* Cancer within 5 years
* Not appropriate for oral antidiabetic agent
* Medication which affect glycemic control
* Disease which affect efficacy and safety of drugs
* Other clinical trial within 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The change of HbA1c | 24weeks

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) | 24 weeks
Postprandial Plasma Glucose (PPG) | 24 weeks
Hypoglycemia | 24 weeks
Body weight | 24 weeks
HbA1c < 7.0% without hypoglycemia | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD,PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Hong AR, Lee J, Ku EJ, Hwangbo Y, Kim KM, Moon JH, Choi SH, Jang HC, Lim S. Comparison of vildagliptin as an add-on therapy and sulfonylurea dose-increasing therapy in patients with inadequately controlled type 2 diabetes using metformin and sulfonylurea (VISUAL study): A randomized trial. Diabetes Res Clin Pract. 2015 Jul;109(1):141-8. doi: 10.1016/j.diabres.2015.04.019. Epub 2015 May 5. PMID 26003889